CLINICAL TRIAL: NCT01114594
Title: Pilot Study of RNA as a Biomarker for Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Type: Observational
Sponsor: The Rogosin Institute (Other)
Collaborators: Rockefeller University (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1003010924
Record Dates: First submitted 2010-04-26; First posted 2010-05-03 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Chronic Kidney Disease; Polycystic Kidney, Autosomal Dominant
Keywords: Chronic Kidney Disease (CKD); Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, monocytes, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PKD: Patients with Autosomal Dominant Polycystic Kidney Disease
- non-PKD CKD: Patients with non-Polycystic Chronic Kidney Disease

SUMMARY:
The aim of this pilot project is to assess the potential of urine micro-RNAs (miRNA) as biomarkers for characterizing patients with autosomal dominant polycystic kidney disease (ADPKD) compared with patients with other causes of chronic kidney disease.

DETAILED DESCRIPTION:
Proteins and small molecules in urine (biomarkers) have been used to probe for kidney and systemic diseases for hundreds of years. Urine reportedly contains a type of molecule called microRNA (miRNAs) that regulate a large number of biological processes. Impaired function of miRNAs is now recognized in an increasing number of disease processes. In the search for new biomarkers, the regulatory function of miRNAs and the relative simplicity and precision of characterizing miRNAs, are potential advantages when compared to traditional biomarkers.

The aim of this pilot project is to assess the potential of urine miRNAs as biomarkers for characterizing patients with autosomal dominant polycystic kidney disease (ADPKD), the most prevalent inherited cause of kidney failure. Individuals with other causes of chronic kidney disease (e.g., diabetes, glomerulonephritis), who are matched for key characteristics (e.g. age, sex, level of kidney function) will serve as the control population. A technique for isolation of miRNAs from urine samples will be tailored for the specific needs of this project. Biochemical and computational analysis of small RNAs from these samples will provide urine miRNA profiles and key variability statistics that will be use to design follow-up projects involving patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject, 18 years of age or older, with diagnosis of ADPKD or non-PKD-CKD
2. If female, not pregnant.
3. Willing and able to understand and sign informed consent

Exclusion Criteria:

1. Presenting with any signs or symptoms of an infectious disease
2. Bacterial infection determined by urine culture
3. Use of systemic steroids within a week prior to screening
4. History, physical, or laboratory findings suggestive of any other medical or psychological condition that would, in the opinion of the Principal Investigator, make the candidate ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 outpatients, 20 patients control
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Identification of micro-RNA Biomarkers Associated with Autosomal Dominant Chronic Kidney Disease | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jon Blumenfeld, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States